CLINICAL TRIAL: NCT06414486
Title: Evaluation of the Effects of Botalys Red Panax Ginseng on Cognitive, Psychological and Emotional Processing in Stressed Adults
Brief Title: Effects of Ginseng on Stress, Emotional and Cognitive Processing
Acronym: GNIZEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Botalys (Industry)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GINZEN
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stress
Keywords: Panax ginseng; Stress; Fatigue; Emotion processing
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Comparative, randomized, placebo-controlled, double-blind, monocentric interventional study in parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement group (Experimental): Participants received orally 1 tablet containing 200mg of Red Panax Ginseng for 4 weeks
  Interventions: Dietary Supplement: Dietary supplement group
- Control group (Placebo Comparator): Participants received orally 1 tablet similar to the test product, containing no active principle for 3 weeks
  Interventions: Other: Placebo group

INTERVENTIONS:
Dietary Supplement: Dietary supplement group — One tablet per day for 3 weeks consumed for subjects randomized in the Dietary supplementation group. This will lead to an intake of 200mg per day of Red Panax Ginseng (corresponding to 22.4mg of ginsenosides and 20.2mg of rare ginsenosides).
  Arms: Dietary supplement group
Other: Placebo group — One tablet per day consumed for 3 weeks for subjects randomized in the Control group. The product is composed of rice flour (50mg) and brown sugar (150mg).
  Arms: Control group

SUMMARY:
This study aims to confirm the positive effect of the Red Panax Ginseng on the cognitive performance and regulation of stress and fatigue in adults with moderate stress level.

DETAILED DESCRIPTION:
This study has been designed as a randomized double-blind placebo-controlled interventional study.

One hundred and fifty participants (aged between 18 and 60), presenting a moderate level of perceived stress, were randomly allocated to the control (placebo) or test (ginseng supplement) group. Participants will be supplemented during 3 weeks with those products. Cognitive performance and emotional processing will be measured with tests and questionnaires before (baseline) and at the end (3 weeks) of the intervention. Fasted blood glucose level will be measured in blood before (baseline) and at the end (3 weeks) of the intervention.

ELIGIBILITY:
Inclusion Criteria:

I.1. Healthy woman or man, aged of 18 to 60 years (inclusive); I.2. With a moderate level of perceived stress (PSS scores ranging from 14 to 26); I.3. Provision of signed and dated informed consent form; I.4. Stated willingness to comply with all study procedures and availability for the duration of the study; I.5. Speaking French.

Exclusion Criteria:

E.1. Subject with severe medical or cognitive problems which, in the opinion of the Principal Investigator, could interfere with the evaluation of the study criteria or with participant safety; E.2. Subject with a coffee consumption of more than 5 cups per day; E.3. Subject consuming drugs and/or with historical drug addiction (<5 years); E.4. Subject with alcohol consumption exceeding 3 glasses of wine per day, or two halves of a beer per day, or one glass of strong alcohol per day; E.5. Subject undergoing medical treatment which, in the opinion of the Principal Investigator, could interfere with cognitive and emotional processing; E.6. Subject with type 1 or type 2 diabetes; E.7. Subject participating in another intervention trial; E.8. Women of childbearing age who are pregnant or breastfeeding or who wish to become pregnant within the next 6 weeks or who are not using an adequate method of contraception (e.g. oral contraception, IUD, abstinence, ...).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
A decrease of stress level | 3 weeks
  Comparison between groups of the adjusted for baseline stress level assessed by the Perceived Stress Scale (PSS)

SECONDARY OUTCOMES:
Evolution of depression state | 3 weeks
  Comparison between groups of the adjusted for baseline of depression state (BDI)
Evolution of anxiety state | 3 weeks
  Comparison between groups of the adjusted for baseline of anxiety state (STAI-S)
Evolution of emotional processing | 3 weeks
  Comparison between groups of the adjusted for baseline of emotional processing assessed by the PANAS
Evolution of fatigue level | 3 weeks
  Comparison between groups of the adjusted for baseline of fatigue level (PIC)
Evolution of attentional performance | 3 weeks
  Comparison between groups of the adjusted for baseline of attentional performance assessed by the Reaction Time and Rapid Visual Information Processing subtests of CANTAB.
Evolution of memory performance | 3 weeks
  Comparison between groups of the adjusted for baseline of memory performance assessed by the Verbal Recognition Memory, Paired Associate Learning and Spatial Span subtests of CANTAB.
Evolution of executive functions performance | 3 weeks
  Comparison between groups of the adjusted for baseline of executive functions performance assessed by the Multitasking Test and One Touch Stockings of Cambridge subtests of CANTAB.
The intervention satisfaction of the volunteer | 3 weeks
  Comparison between groups of the adjusted for baseline of the intervention satisfaction of the volunteer, evaluated by a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Louise Deldicque, Prof, Study Director — Université Catholique de Louvain; Sylvie Copine, Dr, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Center of Investigation in Clinical Nutrition (CICN), Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No